CLINICAL TRIAL: NCT03228901
Title: Exploring the Effects of Oxytocin on Non-verbal Communication
Brief Title: Oxytocin and Non-verbal Communication
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale-NUS College (Other)
Responsible Party: Principal Investigator, Jean Liu, Assistant Professor, Yale-NUS College
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Basic Science
Other Study IDs: IG15-B052
Record Dates: First submitted 2017-07-21; First posted 2017-07-25 (Actual); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Social Interaction
Keywords: Oxytocin; Affiliation
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxytocin (Experimental): 24IU Syntocinon, delivered in a single nose via a nasal spray
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator): Matched nasal spray
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Oxytocin — Administration of the hormone oxytocin
  Other Names: Syntocinon
  Arms: Oxytocin
Drug: Placebos
  Arms: Placebo

SUMMARY:
In this protocol registration, the investigators plan a secondary data analysis of a dataset to explore the effects of intra-nasal oxytocin on the non-verbal expression of affiliation.

DETAILED DESCRIPTION:
Using Liu et al.'s (2012) dataset, the investigators seek to observe whether the administration of oxytocin modifies non-verbal communication with a stranger.

This dataset involves a conversation between two strangers that took place 45 minutes after drug administration. While Liu et al. coded the video for markers of interpersonal distance (physical distance, eye contact, conversational intimacy), the investigators seek to analyse oxytocin's effects on non-verbal communication of affiliative and sexual cues (e.g., smiles, lip puckers). Based on findings that oxytocin's effects depend on context, the investigators will explore these relationships as a function of the conversational context (where participants converse with each other using low-, medium-, and high-intimacy topics, or in an unstructured conversation).

ELIGIBILITY:
Inclusion Criteria:

* healthy

Exclusion Criteria:

* pregnant;
* history of epilepsy, severe depression, severe anxiety, or psychosis;
* smoking more than 15 cigarettes a day;
* addicted to illegal substances.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2007-01 (Actual); Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Non-verbal communication | Measured in the interaction which commenced 45mins after drug administration
  Based on coding the video-recorded interaction between two strangers, using a coding scheme by Gonzaga et al. (for affiliative and sexual cues)

SECONDARY OUTCOMES:
Ratings of the person participants interacted with | Measured following the interaction (which commenced 45 mins after drug administration)
  Positivity or sexual attraction towards the other participant in the conversation (as measured using visual analogue scales based on person perception studies)

CONTACTS AND LOCATIONS:
Locations (1):
- University of New South Wales, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No